CLINICAL TRIAL: NCT06330909
Title: Image-guided Focal Dose Escalation in Patients With Primary Prostate Cancer Treated With Primary External Beam Hypofractionated Stereotactic Radiation Therapy (HypoFocal-SBRT) - a Prospective, Multicenter, Randomized Phase III Study
Brief Title: Image-guided Focal Dose Escalation- Primary pc Treated With Primary External Beam Hypofract.Stereotactic rt
Acronym: HypoF-SBRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. med. Anca-Ligia Grosu, Prof. Dr. med., University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P003103; DRKS00022915 (Other: Deutsches Register Klinische Studien)
Record Dates: First submitted 2023-05-23; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; HypoFocal; HypoFocal-SBRT
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiotherapy, Intensity-Modulated; Radiotherapy, Image-Guided; Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized two arm phase III multicentre trial comparing image-guided focal dose escalation using SBRT in patients with primary PCa treated with primary external beam hypofractionated radiation therapy.
  Patients will be randomized to either arm A (experimental intervention) or arm B (control intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - IMRT/IGRT/SBRT (Experimental): Prostate and seminal vesicles RT with 30 Gy in 6 Gy / fraction; prostate RT with 35 Gy in 7 Gy / fraction including a simultaneous integrated boost (SIB) on the intraprostatic tumour mass (ITM) with 40- 42 Gy in 8 - 8.4 Gy / fraction.
  If the boost volume is ≥10 ml and/ or ≥ 1/3 of the prostate, the SIB on the ITM has to be restrained to 40 Gy in 8 Gy / fraction. SBRT will be performed twice a week, with at least 2 days between two RT fractions, 5 fractions in 3 weeks (technique: IMRT/IGRT/SBRT).
  Interventions: Radiation: Radiotherapy (RT) Arm A - IMRT/IGRT/SBRT
- Arm B - IMRT/IGRT (Active Comparator): Prostate and seminal vesicles RT with 46.4 Gy in 2.32 Gy per fraction, prostate RT with 60 and 62 Gy in 3 and 3.1 Gy per fraction for unfavorable intermediate-risk and high-risk patients, respectively, 20 fractions, 5 fractions /week, (technique: IMRT/IGRT).
  Interventions: Radiation: Radiotherapy (RT) Arm B - IMRT/IGRT

INTERVENTIONS:
Radiation: Radiotherapy (RT) Arm A - IMRT/IGRT/SBRT — technique: IMRT/IGRT/SBRT
  The HypoFocal-SBRT study combines ultra-hypofractionated RT / stereotactic body RT (reduction of treatment time) with a focal RT dose escalation on intraprostatic tumor sides by applying state of the art diagnostic imaging and most modern RT concepts.
  Other Names: Intensity modulated radiotherapy (IMRT); Image guided radiotherapy (IGRT); Stereotactic Body Radiation Therapy (SBRT)
  Arms: Arm A - IMRT/IGRT/SBRT
Radiation: Radiotherapy (RT) Arm B - IMRT/IGRT — technique: IMRT/IGRT
  Moderate hypofractionated RT (MHRT), one option for the curative primary treatment of PCa, which has been proven by several prospective trials and is recommended and carried out worldwide.
  Other Names: Intensity modulated radiotherapy (IMRT); Image guided radiotherapy (IGRT)
  Arms: Arm B - IMRT/IGRT

SUMMARY:
Technical advances in radiotherapy (RT) treatment planning and delivery have substantially changed RT concepts for primary prostate cancer (PCa) by (i) enabling a reduction of treatment time and by (ii) enabling a safe delivery of high RT doses. Several studies proposed a dose-response relationship for patients with primary prostate cancer (PCa) and especially in patients with high-risk features a dose escalation should lead to improved tumor control. In parallel to the improvements in RT techniques, diagnostic imaging techniques like multiparametric magnetic resonance imaging (mpMRI) and positron-emission tomography (PET) evolved and enable an accurate depiction of the intraprostatic tumor mass for the first time. The HypoFocal-SBRT study combines ultra-hypofractionated RT / stereotactic body RT (reduction of treatment time) with a focal RT dose escalation on intraprostatic tumor sides by applying state of the art diagnostic imaging and most modern RT concepts. This novel concept will be compared with moderate hypofractionated RT (MHRT), one option for the curative primary treatment of PCa, which has been proven by several prospective trials and is recommended and carried out worldwide. We suspect an increase in relapse-free survival (RFS) and we will also assess quality of life in order to detect potential changes.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most frequent diagnosed malignancy in male patients in Europe and radiation therapy (RT) is a main treatment option. Conventional RT for patients with primary PCa aims at delivering a homogeneous dose to the entire prostatic gland. However, recent studies proved that modern medical imaging is able to detect accurately the intraprostatic tumour mass (ITM). Consequently, RT concepts for PCa have an imminent need to be rectified in order to individualize the RT strategy by considering the individual tumor localization. In addition, the radiobiological characteristics of the major organs at risk, the rectum and urinary bladder / urethra, as well as of the PCa itself speak for clear advantages of hypofractionated radiation therapy. High-precision stereotactic body radiation therapy (SBRT) significantly shortens the duration of treatment, with clear implications for quality of life and socio-economic aspects.

The aim of this prospective, randomized, multicenter phase III study is the personalization of RT for patients with primary PCa based on individual tumor geometry derived from modern imaging techniques (mpMRI and PSMA-PET/CT). In the experimental (arm A) simultaneous RT dose escalation to the ITM will be performed under strict adherence to the organs at risks' dose constraints by using SBRT (ultra-hypofractionated radiation therapy) in a shorter treatment time (5 fractions vs. 20 fractions). In the control arm (arm B) the entire prostatic gland will receive a homogeneous moderately hypofractionated RT according to the current guidelines. RFS after RT (calculated from randomization) will be assessed as the primary endpoint as well as toxicities and patient reported quality of life as secondary endpoints. For the patients in the experimental arm we expect a significant benefit in relapse free survival (from 80% to 90% at 5 years). The improvement in relapse free survival could increase the metastatic free survival, prostate cancer survival and overall survival in high risk PCa patients. Considering the epidemiological importance of the PCa these results could have a significant socio-economic impact. In parallel a translational research program will address the identification of novel biomarkers/bio-imaging-markers predictive for outcome after RT. Furthermore, involvement of patient representatives includes information about the studies status and contributes to patient empowerment. These aspects will facilitate the evolution from an individualized RT to a personalized RT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate (histological confirmation can be based on tissue taken at any time, but a re-biopsy should be considered if the biopsy is more than 12 months old)
2. Primary localized PCa (cN0 and cM0 in mpMRI and PSMA PET):

   * high- or very high-risk according to NCCN v2.2021 (see 20.3) OR
   * unfavorable intermediate-risk disease according to NCCN v2.2021 (see 20.3)
3. Signed, written informed consent for HypoFocal-SBRT study
4. Age > 18 years
5. Previously conducted PSMA-PET/CT and mpMRI scans or PSMA-PET/MR, fulfilling standard requirements for PCa (see also 6.5)
6. ECOG Performance score 0 or 1
7. IPSS Score ≤15
8. Prostate volume ≤75 ml at RT planning

Exclusion Criteria:

1. Evidence of neuroendocrine tumor cells
2. Prior radiotherapy to the prostate or pelvis
3. Prior radical prostatectomy
4. Prior focal therapy approaches to the prostate
5. Time gap between the beginning of ADT and conduction of mpMRI and PSMA PET scans is >1 month
6. Radiologically suspicious or pathologically confirmed lymph node involvement (cN+) in mpMRI and/or PSMA PET/CT
7. Evidence of metastatic disease (cM+) in mpMRI and/or PSMA PET/CT
8. Evidence of cT4 disease in mpMRI or PSMA PET/CT
9. PSA >30 ng/ml prior to starting ADT
10. Expected patient survival <5 years
11. Bilateral hip prostheses or any other implants/hardware that would introduce substantial CT artefacts
12. Contraindication to undergo a mpMRI scan
13. Prostate surgery (TURP or HOLEP) with a significant tissue cavity or prostate surgery (TURP or HOLEP) within the last 6 months prior to randomization
14. Medical conditions likely to make radiotherapy inadvisable e.g. acute inflammatory bowel disease, hemiplegia or paraplegia
15. Previous malignancy within the last 2 years (except basal cell carcinoma or squamous cell carcinoma of the skin), or if previous malignancy is expected to significantly compromise 5 year survival
16. Any other contraindication to external beam radiotherapy (EBRT) to the pelvis
17. In mpMRI and PSMA PET/CT or PSMA PET/MRI scans no visible tumor
18. Participation in any other interventional clinical trial within the last 30 days before the start of this trial
19. Simultaneous participation in other interventional trials which could interfere with this trial; simultaneous participation in registry and diagnostic trials is allowed
20. Patient without legal capacity who is unable to understand the nature, significance and consequences of the trial;
21. Known or persistent abuse of medication, drugs or alcohol
22. Patients expected to have severe set up problems
23. Dose constraints for organs at risk cannot be adhered to

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival | 7 years
  Primary endpoint is relapse free survival (RFS), defined as time from randomization to relapse or death. Relapse free survival times will be censored at the time see last alive without relapse. Analysis will be conducted after finalization of the study.

SECONDARY OUTCOMES:
Time to local failure after randomization | 7 years
  Time to local failure after randomization. Local recurrences have to be confirmed by biopsy
Metastatic free survival after randomization | 7 years
  Metastatic free survival after randomization (all metastases have to be confirmed by imaging, preferably PSMA-PET/CT or mpMR imaging)
Overall (OS) and prostate cancer specific (PCSS) survival after randomization | 7 years
  Overall (OS) and prostate cancer specific (PCSS) survival after randomization
Time to biochemical failure (phoenix definition) after randomization | 7 years
  Time to biochemical failure (phoenix definition) after randomization
Patient reported acute quality of life (QOL) - Expanded Prostate Index Composite-26 (EPIC-26) | at months 3 and 6 after randomization
  Patient reported acute quality of life (QOL). Acute QOL will be assessed with the Expanded Prostate Index Composite-26 (EPIC-26) Short Form and International Prostate Symptom Score (IPSS) questionnaires at the following time points: before treatment (baseline), last day of treatment, FU visits at months 3 and 6 after randomization
Patient reported late quality of life (QOL) | up to 90 after randomization
  Patient reported late quality of life (QOL). Late QOL will be assessed with the Expanded Prostate Index Composite-26 (EPIC-26) Short Form and International Prostate Symptom Score (IPSS) questionnaires at the following time points: FU visits at months 9,12,15,18 21, 24, 30, 36, 42, 48 and months 54, 60, 66, 72, 78, 84 up to 90 after randomization
Cumulative acute GU and GI toxicities during and up to 3 months after RT using the CTCAEv5.0 criteria | up to 3 months
  Cumulative acute GU and GI toxicities during and up to 3 months after RT using the CTCAEv5.0 criteria
Cumulative Chronic GU and GI toxicities after RT using the CTCAEv5.0 criteria | 7 years
  Cumulative Chronic GU and GI toxicities after RT using the CTCAEv5.0 criteria
Dose constraints and prescription doses / recruited patients | 7 years
  Feasibility and adherence to dose constraints by measuring the ratio between: number of patients with fulfilled dose constraints and prescription doses / recruited patients
Characterization of safety: adverse events | 7 years
  Characterization of safety: adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Anca-Ligia Grosu, Prof., Study Chair — Medical Center- University of Freiburg
Locations (1):
- Medical Center - University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No